CLINICAL TRIAL: NCT00389935
Title: Thalidomide Reduces Arteriovenous Malformation Related Gastrointestinal Bleeding
Acronym: TAG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northport Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Augusta University (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Atul Kumar, US Veterans Affairs Medical Center Northport
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00198
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-07

CONDITIONS: Arteriovenous Malformation; Hereditary Hemorrhagic Telangiectasia; Hematochezia; Melena
Keywords: Gastrointestinal Bleeding; Arteriovenous Malformation; Angiodysplasia; Hereditary Hemorrhagic Telangiectasia; Obscure Bleeding
MeSH Terms: conditions — Arteriovenous Malformations; Telangiectasia, Hereditary Hemorrhagic; Gastrointestinal Hemorrhage; Melena; Angiodysplasia | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: Thalidomide — Thalidomide 50 - 200 mg once at nightime

SUMMARY:
The purpose of this study is to determine whether Thalidomide is effective in the treatment of arteriovenous malformations in the gastrointestinal tract.

DETAILED DESCRIPTION:
Arteriovenous malformations (AVM's) are the commonest vascular abnormalities of the gut. AVM's or Angiodysplasia may be acquired or inherited as in a hereditary hemorrhagic telangiectasia (HHT). Repeated episodes of gastrointestinal bleeding (GIB), especially in the elderly have been attributed to angiodysplasia. Clinically significant GIB may be also seen in up to 40% of HHT patients, usually in the fourth and fifth decades of life. GIB may manifest both as acute major hemorrhage, slow intermittent blood loss or a combination of these findings and patients may be symptomless, present with acute bleeding or iron deficiency anemia. Recurrent hemorrhage and persistent iron-deficiency anemia is common despite supplemental iron therapy and patients require repeated transfusions. Amongst patients with preexisting co-morbidities, repeated bleeding may lead to significant morbidity and mortality. Furthermore, re-bleeding among these patients consumes a disproportionate share of healthcare resources devoted to multiple admissions, repeated endoscopies and blood transfusions. There are no effective treatment options available currently. The purpose of this study is to determine whether Thalidomide is effective in the treatment of arteriovenous malformations in the gastrointestinal tract.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older
* Patient must have had greater than 2 episodes of overt bleeding over last 2 years requiring > 4 units of PRBC for bleeding 20 AVM. AVM's should have been identified at optical/capsule endoscopy or angiography.
* Patients must have adequate hematologic, renal and liver function (i.e. Platelets ≥ 100,000/mm3, Creatinine ≤ 1.7mg/dl, Total Bilirubin ≤ 2.5mg/dl, Transaminases ≤ 4 times above the upper limits of the institutional norm)
* Patients must be able to provide written informed consent. Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods (described in detail under thalidomide drug information section) to avoid conception. Women of child-bearing potential must have a negative pregnancy test prior to treatment on this protocol. Men taking thalidomide must agree to use latex condoms every time they have sex with women since it has been shown that thalidomide is found in semen. All patients must agree to participate in the S.T.E.P.S.® program (System for Thalidomide Education and Prescribing Safety). All patients must be educated under the requirements of the S.T.E.P.S.® program. Patients are required to complete a S.T.E.P.S.® survey and sign and additional consent form indicating that they understand all information provided to them as part of the S.T.E.P.S.® educational counseling.
* Estimated life expectancy must be greater than 2 months.

Exclusion Criteria:

* Pregnant and/ or lactating female
* Personal history of thromboembolic disease
* History of seizure activity
* History of neoplasm except basal cell carcinoma in-situ
* History of severe neuropathies
* Women of child bearing potential
* Inability to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-10; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Blood Transfusion requirements | 6 months

SECONDARY OUTCOMES:
Hemoglobin overall complication rate Constipation Neuropathy | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Atul Kumar, MD, Principal Investigator — Northport VAMC; James Gossage, MD, Principal Investigator — Augusta University
Locations (3):
- United States (3):
  - Medical College of Georgia, Augusta, Georgia
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Northport VAMC, Northport, New York